CLINICAL TRIAL: NCT05196490
Title: Analyzing the Effect of Sodium Bicarbonate and Glycine Air Polishing on Tooth Surfaces With Two Different Imaging Methods
Brief Title: Analyzing the Effect of Air Polishing on Tooth Surfaces With Two Imaging Methods
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Vecihe Merve Balta Uysal, Lecturer, Kocaeli University
Other Study IDs: KOU GOKAEK 2020/08.07
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Dental Plaque
Keywords: computer-aided design; X-Ray microtomography; sodium bicarbonate; glycine; air abrasion
MeSH Terms: conditions — Dental Plaque | interventions — X-Ray Microtomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Micro-CT: Samples were scanned before and after air polishing with a high-resolution micro-CT device. The scanning conditions were 100 kVp; 100-mA, 0.5-mm Al/Cu filter; 13.1-μm pixel size; and rotation at 0.2 steps. According to the manufacturer's instructions, each sample was rotated 360°. The mean scanning time was around 1hour.
  Interventions: Device: Micro-CT
- CAD/CAM: The teeth surfaces were digitalized before and after air polishing with an intraoral scanner. The mean scanning time was around 10 second. The virtual images of the scanned teeth were saved in stereolithography (STL) format.
  Interventions: Device: CAD/CAM

INTERVENTIONS:
Device: Micro-CT — Micro computed tomography (micro-CT) is an imaging method in which cross-sectional images are obtained and these images are transferred to the computer through specific software, processed and stored.
  Groups: Micro-CT
Device: CAD/CAM — CAD/CAM (computer aided design-computer aided manufacturing) is a production method that is frequently used in many areas of technology. These systems are composed of a data acquisition unit, software for designing virtual restoration, and a computerized milling device.
  Groups: CAD/CAM

SUMMARY:
Micro-CT is a non-destructive imaging method with high resolution and allows to examine all tooth structures individually. Pre- and post-application images obtained by micro-CT can be superimposed and differences can be precisely detected. Intraoral scanners in CAD/CAM systems also provide non-destructive image scanning. CAD/CAM are systems that are widely used in dentistry today. Access to the device is easier than micro-CT. This study was focused on to compare two different imaging methods by assessing changes caused by sodium bicarbonate and glycine air polishing on the tooth surfaces.

DETAILED DESCRIPTION:
The patients were recruited from individuals seeking periodontal and/or dental treatment at Kocaeli University, Faculty of Dentistry. The teeth samples were collected from the participants who have a single-rooted tooth with the gingival recession on all surfaces and need to be extracted. All patients who met the criteria were informed about the study. Patients who gave written informed consent were included. Before the teeth extractions, root surfaces were marked with a bur at the level of the gingival margin. Extractions were performed under local anesthesia with 2% xylocaine adrenalin. Fourteen single root extracted teeth were included into the study. The crown and exposed root surface were air polished using glycine and sodium bicarbonate powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree.

Samples were scanned before and after air polishing with a high-resolution micro-CT device. The scanning conditions were 100 kVp; 100-mA, 0.5-mm Al/Cu filter; 13.1-μm pixel size; and rotation at 0.2 steps. According to the manufacturer's instructions, each sample was rotated 360°. The mean scanning time was around 1hour. The teeth surfaces were digitalized before and after air polishing with an intraoral scanner. The mean scanning time was around 10 second. The virtual images of the scanned teeth were saved in stereolithography (STL) format. The defect volume was estimated.

The data were analyzed using commercially available statistical analysis software. Descriptive statistics that were used to analyze the results included the mean, standard deviation, median, minimum, and maximum. Mann-Whitney U test was performed to compare differences between two independent variables. Wilcoxon test was used to compare differences between two dependent variables. P-values less than 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Being older than age of 18, Willing to participate the study, To have a single rooted tooth with gingival recession on all surfaces and need to be extracted, The tooth has to be free of caries, defects and restorations.

Exclusion Criteria:

Have history of infectious diseases like Hepatitis and/or HIV (+).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients were recruited from individuals seeking periodontal and/or dental treatment at Kocaeli University, Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Defect volume | 5 second
  The teeth were divided into two groups, the crown and exposed root surface were air polished using glycine and sodium bicarbonate powders at instrumentation time of 5s, combinations of medium and maximum power and medium water settings, distance of 5mm and angulation of 60 degree. Samples were scanned in a micro-computed tomography (micro-CT) and CAD/CAM at baseline and then after powder treatment and the defect volume was estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Faculty of Dentistry, Kocaeli, Turkey (Türkiye)